CLINICAL TRIAL: NCT05856201
Title: Laparoscopic Supracervical Hysterectomy With Cervicosacropexy and Vaginally Assisted NOTES Hysterectomy With Uterosacral Ligament Suspension (Shull Technique): a Randomized Multicentric Prospective Comparison Trial
Brief Title: Laparoscopic Sacropexy and Vaginal Natural Orifice Transluminal Endoscopic Surgery Shull Suspension Comparison Trial
Acronym: V-PULSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Tommaso Simoncini, Principal Investigator, Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V-PULSE study
Record Dates: First submitted 2023-04-20; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: We will perform a interventional, no profit, prospective, randomized 1:1 multicentre, controlled trial with participating tertiary referral hospital centers in Italy, to compare the laparoscopic cervicosacropexy (CSP) and Shull technique via V-NOTES (VNS) in the management of apical prolapse.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The 6-week examination and review will be performed by the surgeon with all study data and future visits completed by blinded co-authors (Different surgeon or Urogynecology fellows) who will be unaware of group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic cervicosacropexy (CSP) (Active Comparator)
  Interventions: Procedure: Laparoscopic cervicosacropexy
- Shull technique via V-NOTES (VNS) (Active Comparator)
  Interventions: Procedure: Shull technique via V-NOTES

INTERVENTIONS:
Procedure: Laparoscopic cervicosacropexy — The first step consists of a supracervical hysterectomy with morcellation. Anterior and posterior dissection of the vesicovaginal and rectovaginal space. Placing a flexible blade or a Breisky blade in the vagina which is manipulated by the assistant in order to improve exposure of the tissue planes. The retroperitoneum will then be opened from sacral promontory to cervix with the incision just medial to the uterosacral ligament. A low-weight preshaped Y-shaped polypropylene mesh will be secured to the anterior and posterior vagina with four to six separated absorbable 2.0 polyglactin sutures and two nonabsorbable 2.0 prolene sutures can be placed at the level of the remaining cervix. The mesh will be attached to the sacral promontory using two or three nonabsorbable monofilament 2.0 prolene suture. The retroperitoneal space will be closed with continuous 2.0 polyglactin suture or barbed 2.0 absorbable suture material.
  Arms: laparoscopic cervicosacropexy (CSP)
Procedure: Shull technique via V-NOTES — Using a cold-bladed scalpel, pericervical colpotomy and subsequent opening of the Douglas and vesico-uterine space is performed. The following step is forcipressure and section of uterosacral ligaments bilaterally with cold blade scissors and ligation in Polysorb 0. A v-PATH® wall retractor is placed, after insertion of three trocars. Total hysterectomy is then performed by standard V-NOTES technique. After transperitoneal visualization of the ureters bilaterally, the peritoneum is incised between the ureters and the uterosacral ligaments, which are thus bilaterally isolated, and three points in polydioxanone 2/0 are placed per side. The v-PATH wall retractor is then removed. Finally the suspension of the vaginal vault at the uterosacral ligaments is made according to Shull technique. Eventual fascial corrections of concomitant anterior or posterior defects will be associated if needed.
  Arms: Shull technique via V-NOTES (VNS)

SUMMARY:
This is a prospective, randomized multicenter study whose objective is to compare two surgical techniques routinely used at our center for the correction of pelvic organ prolapse (laparoscopic cervicosacropexis versus colposuspension sec. Shull using v-NOTES).

DETAILED DESCRIPTION:
patients with pelvic organ prolapse with a stage greater than or equal to stage 2 for the apical compartment who are candidates for surgical correction will be randomized and assigned to one of two treatment groups. The aim is to compare the anatomical, surgical and anesthesiological outcomes between these two surgical techniques, both of which are commonly used in clinical practice for the correction of this type of prolapse.

ELIGIBILITY:
Inclusion Criteria:

* consecutive women referred to one of the participating centers with symptomatic stage 2 or greater (point C≥ -1 pelvic organ prolapse quantification POP-Q) apical prolapse (uterovaginal) with or without anterior and posterior compartment prolapse will be eligible for inclusion (Criteria for which patients in clinical practice are candidates for one of the two interventions under study)

Exclusion Criteria:

* age <18 years, BMI > 30,
* previous hysterectomy,
* inability to comprehend questionnaires, to give informed consent and to return for review,
* unable to undergo general anesthesia,
* prior laparoscopic prolapse repair or vaginal mesh prolapse procedure,
* desire for future pregnancy or current pregnancy diagnosis
* severe respiratory comorbidity,
* ASA III patients,
* need for concomitant anti-incontinence procedure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
operating time | intraoperative
  from skin/vaginal incision to end of skin/vaginal suture
post-operative pain | at 4 hours post-operative
  VAS (visual analogic scale, from 0 (minimum), to 10 (maximum pain))
post-operative pain | at 8 hours post-operative
  VAS (visual analogic scale, from 0 (minimum), to 10 (maximum pain))
post-operative pain | at 1 month post-operative
  VAS (visual analogic scale, from 0 (minimum), to 10 (maximum pain))
post-operative pain | at 12 hours post-operative
  VAS (visual analogic scale, from 0 (minimum), to 10 (maximum pain))
time to mobilization with standing | immediately post-operative
  Time it takes the patient to mobilize to standing independently
hospital stay | immediately post-operative
  hours of post-operative stay
patient satisfaction | at 6 weeks
  assessed by P-QoL (prolapse quality of life) validated questionnaire
patient satisfaction | at 3 months
  assessed by P-QoL validated questionnaire
patient satisfaction | at 6 weeks
  assessed by PGI-I (patient global impression of improvement) validated questionnaires
patient satisfaction | at 3 months
  assessed by PGI-I validated questionnaires
patient satisfaction | at 6 weeks
  assessed by validated questionnaires (VAS, visual analogic scale from 0 to 10)
patient satisfaction | at 3 months
  assessed by validated questionnaires (VAS, visual analogic scale from 0 to 10)
sexual function | at 6 weeks
  assessed by FSFI (female sexual function index) questionnaire
sexual function | at 3 months
  assessed by FSFI questionnaire
sexual function | at 6 weeks
  assessed by TVL (total vaginal lenght) measure
sexual function | 3 months
  assessed by TVL measure
recurrence of prolapse in apical compartment | at 6 weeks and 3 months;
  POP-Q (Pelvic Organ Prolapse Quantification system) C point measure
recurrence of prolapse in apical compartment | at 6 weeks
  POP-Q (Pelvic Organ Prolapse Quantification system) C point measure
recurrence of prolapse in the anterior and posterior compartments when present | at 3 months;
postoperative complications | from surgery to 3 motnhs follow.up
  assessed using Clavien-Dindo classification
anesthesiological parameters | intraoperative
  End tidal CO2 (carbon dioxide) assessement
anesthesiological parameters | intraoperative
  SpO2 (oxygen saturation) assessement
anesthesiological parameters | intraoperative
  blood pressure assessement (measured in mmHg)
anesthesiological parameters | intraoperative
  intraoperative blood loss assessement (measured in milliliters)
anesthesiological parameters | intraoperative
  degrees of Trendelemburg assessement

IPD SHARING:
Plan to Share IPD: No